CLINICAL TRIAL: NCT04559841
Title: Regenerative Surgical Treatment of Peri-implantitis Using Nanobone With or Without Simvastatin: A 6-month Randomized Controlled Clinical Trial
Brief Title: Regenerative Surgical Treatment of Peri-implantitis Using Nanobone With or Without Simvastatin
Acronym: RAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reham Lotfy Aggour (Other)
Collaborators: October 6 University (Other)
Responsible Party: Sponsor-Investigator, Reham Lotfy Aggour, Associate professor of Oral Medicine, diagnosis & Periodontology, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (IEC)/15-2017
Record Dates: First submitted 2020-09-07; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Peri-Implantitis
Keywords: dental implant; peri-implantitis; surgical treatment
MeSH Terms: conditions — Peri-Implantitis | interventions — Bone Substitutes; NanoBone; Simvastatin

STUDY DESIGN:
Intervention Model Description: single-center, parallel group, 6 month randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: A single examiner blinded to the treatment assignment was responsible for evaluating the clinical parameters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bone substitute; NanoBone® (group 1, control group) (Active Comparator): a synthetic bone substitute consisting of nanocrystalline hydroxyapatite and silica fabricated in a sol-gel process.
  Interventions: Other: bone substitute; NanoBone®
- simvastatin + NanoBone (group 2, test group) (Experimental): medications used to treat hypercholesterolemia
  Interventions: Other: bone substitute; NanoBone®

INTERVENTIONS:
Other: bone substitute; NanoBone® — surgical treatment of peri-implantitis using a regenerative surgical protocol utilizing NanoBone (NB) synthetic bone graft with or without simvastatin.
  Other Names: simvastatin

SUMMARY:
The aim of this study was to evaluate the effect of using a synthetic bone substitute with or without simvastatin on regenerative surgical treatment of bone defects associated with peri-implantitis in a 6- months randomized controlled clinical trial.

A total of 30 patients diagnosed with peri-implantitis were randomly assigned to one of two surgical treatment groups (group I: synthetic bone substitute (NanoBone), group II: NanoBone with simvastatin). Clinical measurements included probing pocket depth (PPD), clinical attachment level (CAL), plaque index (PI), modified sulcus bleeding index (mSBI) and mucosal recession (MR). Radiographic bone fill was evaluated at baseline and after 6- months.

DETAILED DESCRIPTION:
The study was designed as a prospective single-center, parallel group, 6 month randomized clinical trial evaluating the effect of a bone substitute; NanoBone® (Artoss GmbH, Rostock, Germany) (group 1, control group) compared to the same bone substitute with simvastatin (Corvast 80 mg, Egyphar, Egypt) (group 2, test group) for RST of peri-implantitis. A total of 30 patients suffering from peri-implantitis who needed regenerative treatment of at least one peri-implant bone defect were selected and only one implant per patient (the most severe) was evaluated in the treatment groups. The criteria for diagnosing peri-implantitis is based on the consensus report of the eighth European Workshop on Periodontology [34] ; the presence of a peri-implant marginal bone loss ≥2 mm based on baseline periapical radiographs after delivery of the final restoration and bleeding on probing (BOP) and/or suppuration with or without concomitant deepening of peri-implant pockets.

Clinical and radiographic evaluation were conducted at baseline and 6 months postoperatively. Grouping was done using a random number table generated by a third party. They were numbered according to the order of enrolment and assigned to group I or group II. The grouping results were sealed in an opaque envelope and kept by an independent third party. For each patient, cards opened immediately before the surgical procedures. Treatment assignment in each patient was registered by the clinician who assisted in the operations and kept concealed until the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years,
2. having at least one implant demonstrating bone defect ≥3 mm, which presented a probing depth of ≥5 mm with BOP and/or suppuration, implants had to be in function for >12 months,
3. no implant mobility and no evidence of occlusal overload,
4. no evidence of occlusal overload
5. presence of at least 2 mm of keratinized attached mucosa .

Exclusion Criteria:

1. serious systemic diseases, medications or conditions that would contraindicate periodontal surgery and compromise wound healing,
2. history of taking systemic antibiotic during the past 3 months,
3. smoking,
4. pregnant or lactating females,
5. implants previously augmented with bone substitute or placed in grafted bone,
6. implants previously treated for peri-implantitis,
7. a mobile implant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | 6 months
  Clinical attachment level (CAL) defined as probing pocket depth + mucosal recession

SECONDARY OUTCOMES:
probing pocket depth | 6 months
  measured as the distance from the mucosal margin to the base of the deepest pocket of the implant
plaque index (PI) | 6 months
  marked with a score from 0 to 3. Grade 0: no plaque; Grade 1: plaques could be found on the surface of the implant after scratching with the probe tip gently; Grade 2: plaque could be seen by the naked eye; and Grade 3: a large amount of plaques could be seen
Bleeding on probing (BoP) | 6 months
  modified sulcus bleeding index (mSBI) . This index scores the bleeding on a zero to three scale, where 0: no bleeding, 1: isolated bleeding spots, 2: blood forms a confluent red line and 3: heavy or profuse bleeding.
Mucosal recession (MR) | 6 months
  measured as the distance from the mucosal margin and the implant abutment interface
The change in bone level (BL) | 6 months
  the distance (mm) between the implant shoulder and the bottom of the defect

CONTACTS AND LOCATIONS:
Overall Officials: Reham Aggour, Dr, Study Director — Oral Medicine & Periodontology department
Locations (1):
- October 6 University, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided